CLINICAL TRIAL: NCT02663388
Title: Influence of Vitamins Status on Severe Obesity Related Complications
Brief Title: Epigenetic Mechanisms and Severe Obesity (Biological Tissue Collection)
Acronym: OBESEPI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Lorraine (Other)
Collaborators: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Laurent Brunaud, Pr Laurent BRUNAUD, MD, PhD, University of Lorraine
Other Study IDs: 2015-A01175-44
Record Dates: First submitted 2016-01-11; First posted 2016-01-26 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Obesity; Diabetes; Metabolic Diseases; Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Metabolic Diseases; Non-alcoholic Fatty Liver Disease | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — blood, liver, fat tissue (subcutaneous, visceral, mesenteric), small bowell, feces

INTERVENTIONS:
Procedure: gastric bypass, sleeve, gastric banding

SUMMARY:
The purpose of this study was to evaluate the role of vitamin status and epigenetic mechanisms on severe obesity related-complications.

ELIGIBILITY:
Inclusion Criteria:

* indication for bariatric surgery with BMI > 35 kg/m2

Exclusion Criteria:

* unable to receive clear information
* refusal to sign the consent form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who undergo bariatric surgery following french national guidelines (HAS 2009)
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2016-01; Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of folate mediated one-carbon metabolic pathway parameters (Folates, Vitamin B12, Methionine, Homocysteine) on severe obesity-related complications before and after bariatric surgery | 10 years

SECONDARY OUTCOMES:
Evaluation of DNA Methylation on severe obesity-related complications before and after bariatric surgery | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: laurent BRUNAUD, MD, PhD, Principal Investigator — University of Lorraine, CHU Nancy
Locations (1):
- University of Lorraine, CHU Nancy, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Derived] Antoine D, Li Z, Quilliot D, Sirveaux MA, Meyre D, Mangeon A, Brunaud L, Gueant JL, Gueant-Rodriguez RM. Medium term post-bariatric surgery deficit of vitamin B12 is predicted by deficit at time of surgery. Clin Nutr. 2021 Jan;40(1):87-93. doi: 10.1016/j.clnu.2020.04.029. Epub 2020 Apr 25. PMID 32444241
- [Derived] Li Z, Gueant-Rodriguez RM, Quilliot D, Sirveaux MA, Meyre D, Gueant JL, Brunaud L. Folate and vitamin B12 status is associated with insulin resistance and metabolic syndrome in morbid obesity. Clin Nutr. 2018 Oct;37(5):1700-1706. doi: 10.1016/j.clnu.2017.07.008. Epub 2017 Jul 24. PMID 28780990